CLINICAL TRIAL: NCT00428376
Title: Clinical Trial of Building Block Distribution in Children
Brief Title: Does Block Play Improve Language Acquisition: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Megablocks (Unknown)
Responsible Party: Dmitri Christakis, MD, MPH, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 05-0636-01
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Healthy

INTERVENTIONS:
Device: Building Blocks

SUMMARY:
This is a randomized controlled trial of distributing blocks to children ages 1.5 -2.5 years of age to see if language acquisition improves.

DETAILED DESCRIPTION:
Children in age group are randomized to get two sets of blocks or not. Outcomes include language development assessed using the Macarthur Bates CDI 6 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* healthy children

Exclusion Criteria:

* developmental delay, non-English

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Macarthur Bates Language Inventory

SECONDARY OUTCOMES:
TV viewing
Block play

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Christakis, MD MPH, Principal Investigator — University of Washington